CLINICAL TRIAL: NCT05257603
Title: Assessing the Feasibility of a New Prevention to Reduce Alcohol-related Sexual Revictimization of College Women
Brief Title: Prevention of Alcohol-related Sexual Revictimization in College
Acronym: RPCW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kathleen A Parks Marsh, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 86140; R34AA026910-01A1 (NIH)
Record Dates: First submitted 2022-02-08; First posted 2022-02-25 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Sexual Assault
Keywords: Intervention Study; Alcohol Drinking in College
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Intervention Model Description: Half of participants will be assigned to the intervention (RPCW) condition designed to reduce hazardous drinking and increase awareness of risk cues for sexual assault and implementation of safe drinking and dating behaviors. Half of participants will be assigned to the Health education control designed to control for time and attention.
Who Masked: Participant
Masking Description: Participants are not told the outcomes the investigators are seeking to reduce, but are told participants are assigned to either a Health and Lifestyle intervention (Health Education control) or Managing High Risk intervention (RPCW).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revictimization Prevention for College Women (RPCW) (Experimental): Active intervention that includes information to reduce hazardous drinking and increase sexual assault risk perception.
  Interventions: Behavioral: RPCW
- Health Education Control (HEC) (Active Comparator): Time and attention control.
  Interventions: Behavioral: HEC

INTERVENTIONS:
Behavioral: RPCW — Psychosocial intervention that includes two in-person group sessions two weeks apart and two on-line units during the intervening two weeks. Behavioral training, educational materials, discussions and videos, as well as interactive online materials are included to increase awareness of sexual assault cues, dating and drinking protective behavioral strategies, barriers to defending oneself, and saying no to hazardous drinking and sexual advances.
  Arms: Revictimization Prevention for College Women (RPCW)
Behavioral: HEC — Health Education time and attention control that includes two in-person sessions two weeks apart and two on-line units during the intervening two weeks. The in-person sessions cover stress management and sleep, while the online units cover nutrition and physical activity. The in-person and online sessions are designed to foster discussion and be interactive.
  Arms: Health Education Control (HEC)

SUMMARY:
This pilot randomized controlled trial (RCT) is designed to test a new intervention designed to reduce college women's risk for sexual revictimization (SRV). The intervention targets women with a history of sexual assault (SA) and recent hazardous drinking (HD), as these women are at highest risk for SRV. The primary goals of the intervention are to decrease women's HD, improve their ability to perceive cues that signal risk for SRV, and strengthen their behavioral skills in situations associated with an increased risk for SRV. The intervention, Revictimization Prevention for College Women (RPCW) is a multi-modal intervention that includes two on-line interactive education modules and two in-person group skills-based training sessions that focus on problem solving training and behavioral rehearsal. The pilot RCT of the RPCW intervention will include 96 college women with follow-up assessments at 3- and 6-months post intervention. Women will be randomly assigned to either the RPCW intervention or to a Health Education Control (HEC) condition. The pilot RCT will be used to establish the feasibility of recruitment, the acceptability and safety of the RPCW intervention, and provide initial efficacy data that will assist in power calculations for a Stage II efficacy trial. The investigators hypothesize that women in RPCW intervention will report fewer days of hazardous drinking and improved perception of sexual assault risk cues compared with participants in the HEC condition. In addition, women in the RPCW intervention will report increased knowledge of safe dating practices and protective behavioral (drinking) strategies compared with participants in the HEC condition. Finally, women in the RPCW intervention will report lower rates of SRV as compared with participants in the HEC condition at the 6-month post-intervention follow-up.

DETAILED DESCRIPTION:
The investigators will be conducting a Stage 1b randomized controlled trial of a newly developed preventive intervention to reduce sexual revictimization of college women. The preventive intervention, Revictimization Prevention for College Women (RPCW), is designed to reduce sexual revictimization by reducing women's hazardous drinking, and increasing their awareness of protective dating and drinking behavioral strategies, as well as their awareness of risk cues for sexual assault during social situations. The intervention involves two in-person group skills-based training sessions held one week apart and two online interactive educational sessions designed for completion between the in-person sessions. During the pilot RCT, the active intervention (RPCW) will be compared to a time and attention Health Education Control.

The first group session of the RPCW involves viewing 4 cue recognition training videos and participating in an Interventionist lead discussion intended to highlight sexual assault risk cues in each of the videos. After the session, each participant will then complete two interactive, online learning module focused on safe drinking and safe dating. The second group session will occur one week after the first and is designed to elicit feedback on the drinking and dating learning modules (e.g., length, ease of use, engagement, interest). The training videos will be viewed again individually and participants will engage in behavioral skills rehearsal of appropriate responses in paired role plays with feedback from the Interventionist and a group discussion about the emotional barriers to engaging in appropriate dating and drinking safety behaviors (e.g., "I feel bad for the guy", "He might get really mad, "I might miss out on being with a great guy") and strategies for overcoming these barriers. Adaptive emotion regulation strategies will be used such as cognitive reappraisal, distress tolerance, mindfulness of current emotions, acceptance, and problem solving. Immediately following this session, participants will be asked to complete a post-intervention survey, including feedback on the intervention content and process. Following the in-person RPCW sessions, a debriefing will occur to ensure that women have an opportunity to discuss any emotional discomfort or distress with the interventionist. Follow-up surveys will be administered again at 3- and 6-months post intervention. The Health education control (HEC) is a time and attention control and was developed in parallel with the RPCW. The two in-person sessions and two online units of the HEC condition will impart health information that is relevant and engaging for college women but does not directly address heavy drinking or sexual assault risk. It is intended to control for nonspecific intervention factors related to health behavior change. This 4-session active control condition will begin with an in-person session focused on stress management. The second in-person session focuses on sleep hygiene. The two online, interactive modules address nutrition on college campuses and physical exercise. These two modules are similar in format to the drinking and dating safety modules provided in the RPCW. To ensure that HEC participants receive SA risk reduction and HD reduction information, the participants will have the opportunity to receive the RPCW intervention following the 6-month follow-up assessment, if the participants choose to do so.

All participants will participate in the intervention over one week. The participants will attend two in-person group intervention sessions one week apart, and complete their two on-line units during the intervening week. The participants will be asked to complete a baseline survey prior to their first in-person session, a post-intervention session following their second in-person session and two follow-up on-line assessment surveys at 3 months and 6 months post intervention.

The investigators have three specific hypotheses for the RCT:

Hypothesis a: Participants in the RPCW intervention will report fewer days of hazardous drinking and improved perception of SRV risk cues on the video risk perception measure (primary outcomes) as compared with participants in the HEC condition.

Hypothesis b: Participants in the RPCW intervention will report increased knowledge of safe dating practices and protective behavioral (drinking) strategies (secondary outcomes) compared with participants in the HEC condition.

Hypothesis c: Participants in the RPCW intervention will report lower rates of SRV as compared with participants in the HEC condition at 6-month post-intervention follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18-22 years of age
* Current first- or second-year female student at the college
* Able to comprehend the study protocol, consent form and provide written consent
* Had a prior SA experienced since the age of 14 years (i.e., adolescent or young adult)
* Engaged in hazardous drinking in the past month (i.e., ≥ 4 drinks 1 or more times in past 30 days).

Exclusion Criteria:

* Major mental illness as indicated by: (a) severe level of depressive symptoms as assessed by the Beck Depression Inventory-II or a self-reported diagnosis of: (b) Schizophrenia, (c) Bipolar Disorder
* Report experiencing homicidal or suicidal ideation
* Unable to commit to attending 2 weekly in-person group sessions
* No access to a computer to complete the on-line intervention modules.

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — cis-gender female or non-binary, but must be sexually attracted to men.
Enrollment: 72 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ParksMarsh A Kathleen, PhD, Principal Investigator — SUNY Buffalo
Locations (1):
- State University of New York Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared upon request to the researchers in writing.
Supporting Information: Study Protocol, CSR
Time Frame: All information will be shared 6 months after findings are published.
Access Criteria: Information will be available by contacting the PI of the study at kparks@buffalo.edu

REFERENCES:
- [Background] Gratz KL, Roemer, L. Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment. 2004; 26(1): 41-54.
- [Background] Koss MP, Gidycz CA, Wisniewski N. The scope of rape: incidence and prevalence of sexual aggression and victimization in a national sample of higher education students. J Consult Clin Psychol. 1987 Apr;55(2):162-70. doi: 10.1037//0022-006x.55.2.162. No abstract available. PMID 3494755
- [Background] Martens MP, Ferrier AG, Sheehy MJ, Corbett K, Anderson DA, Simmons A. Development of the Protective Behavioral Strategies Survey. J Stud Alcohol. 2005 Sep;66(5):698-705. doi: 10.15288/jsa.2005.66.698. PMID 16329461
- [Background] Martens MP, Pederson ER, Labrie JW, Ferrier AG, Cimini MD. Measuring alcohol-related protective behavioral strategies among college students: further examination of the Protective Behavioral Strategies Scale. Psychol Addict Behav. 2007 Sep;21(3):307-15. doi: 10.1037/0893-164X.21.3.307. PMID 17874881
- [Background] Parks KA, Levonyan-Radloff K, Dearing RL, Hequembourg A, Testa M. Development and Validation of a Video Measure for Assessing Women's Risk Perception for Alcohol-Related Sexual Assault. Psychol Violence. 2016 Oct;6(4):573-585. doi: 10.1037/a0039846. PMID 27747131
- [Background] Lavender JM, Tull MT, DiLillo D, Messman-Moore T, Gratz KL. Development and Validation of a State-Based Measure of Emotion Dysregulation. Assessment. 2017 Mar;24(2):197-209. doi: 10.1177/1073191115601218. Epub 2016 Jul 27. PMID 26297011
- [Background] Hanson KA, Gidycz CA. Evaluation of a sexual assault prevention program. J Consult Clin Psychol. 1993 Dec;61(6):1046-52. doi: 10.1037//0022-006x.61.6.1046. PMID 8113482

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via email and through fliers posted on campus. Cohort 1 was recruited and screened for eligibility over the telephone between February 2, 2022 and April 19, 2022. Cohort 2 was recruited and screened for eligibility over the telephone between September 7, 2022 and April 11, 2023.
Pre-assignment Details: Participants who were screened as eligible, provided informed consent to participate, were assigned to condition and completed the first in-person session of the study protocol were considered to have entered the controlled trial. Therefore, participants could have been eligible, consented and assigned to condition, but if they did not complete the baseline measure or attend the first in-person session, they would not have been considered a participant in the clinical trial.
Groups:
- Revictimization Prevention for College Women (RPCW): Active intervention that includes information to reduce hazardous drinking and increase sexual assault risk perception.
  RPCW: Psychosocial intervention that includes two in-person group sessions two weeks apart (Cohort 1) or one week apart (Cohort 2) with two on-line units during the intervening two weeks. Behavioral training, educational materials, discussions and videos, as well as interactive online materials are included to increase awareness of sexual assault cues, dating and drinking protective behavioral strategies, barriers to defending oneself, and saying no to hazardous drinking and sexual advances.
- Health Education Control (HEC): Time and attention control.
  HEC: Health Education time and attention control that includes two in-person sessions two weeks apart (Cohort 1) or one week apart (Cohort 2) with two on-line units during the intervening two weeks. The in-person sessions cover stress management and sleep, while the online units cover nutrition and physical activity. The in-person and online sessions are designed to foster discussion and be interactive.
Period: Overall Study
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
Started | 37 | 35
Cohort 1: Completers of Two-week Protocol (Completed both in-person group sessions and the two on-line units during the two weeks designated for cohort 1.) | 8 | 5
Cohort 2: Completers of One-week Protocol (Completed both in-person group sessions and the two on-line units during the one week designated for cohort 2.) | 22 | 25
Completed Partial Protocol. (Completed some of the components of the intervention or control.) | 7 | 5
Post-Intervention Survey | 33 | 29
3-Month Follow-up Survey | 32 | 26
Completed One or More Follow-up Visits | 35 | 33
6-Month Follow-up Survey | 29 | 22
Completed (This was an intent to treat sample so all participants who began the trial were considered to have completed for analysis purposes.) | 37 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC) | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 35 | 72
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  cis-gender female | 37 | 35 | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 37 | 35 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 10 | 22
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 35 | 72

OUTCOME MEASURES:

1. Primary Outcome: Days Per Month Hazardous Drinking
Description: A hazardous drinking day is defined as consumption of 4 or more drinks on a given day/drinking occasion during a month. Average number of hazardous drinking days per month will be assessed at each assessment interval.
Time Frame: Baseline to post-intervention (approximately 1 to 2-weeks); Post-intervention to 3-month follow up; 3- to 6-month follow up
Population: Change in number of participants analyzed in different rows indicates the number of participants who completed each of the follow-up measurements. In other words, it indicates the attrition from follow-up after completing the intervention. This was an intent to treat analysis, so all participants were included.
Measure: Mean (Standard Deviation); unit: Days per Month Hazardous Drinking
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
Number analyzed (Participants) | 37 | 35
Days per Month Hazardous Drinking
  Baseline | 7.54 (6.55) | 10.40 (11.51)
  Post-Intervention: number analyzed (Participants) | 33 | 30
  Post-Intervention | 1.97 (2.80) | 1.53 (1.91)
  3-Month Follow Up: number analyzed (Participants) | 32 | 27
  3-Month Follow Up | 3.72 (4.24) | 3.52 (6.30)
  6-Month Follow Up: number analyzed (Participants) | 27 | 19
  6-Month Follow Up | 4.89 (6.85) | 3.89 (4.87)
Statistical Analysis 1: Comparison: Revictimization Prevention for College Women (RPCW) vs Health Education Control (HEC); Test type: Other; p < 0.99, ANOVA; Mean Difference (Net) = 4.82, 95% CI 2-sided [3.24 to 5.72], Standard Error of Mean 0.615

2. Primary Outcome: Severe Sexual Assault (Revictimization)
Description: Any form of severe sexual aggression greater than unwanted contact/touching as measured by the modified sexual experiences survey (Koss et al., 1987) since the intervention ended.
Time Frame: At 6-month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
Number analyzed (Participants) | 37 | 35
Participants
  Sexually Assaulted | 5 | 7
  Not Sexually Assaulted | 32 | 28
Statistical Analysis 1: Comparison: Revictimization Prevention for College Women (RPCW) vs Health Education Control (HEC); Test type: Other; p < .29, Chi-squared

3. Primary Outcome: Mean Number of Key Presses When Watching Risk Video
Description: Improved ability to perceive sexual assault risk was assessed by participants' responses while watching the high- risk video from the Video Vignette Risk Perception Measure (Parks et al., 2016). Increased perception of risk was measured by an increase in the number of times an individual indicated concern when watching the video as measured by pressing a specified key (e.g., "b") on the computer keyboard in response to feeling concerned or uncomfortable while watching the social interaction in the video. An improvement in risk perception was indicated by a higher mean number of key presses. Therefore, a higher mean number of key presses at time 2 compared to time 1 would indicate improved risk perception.
Time Frame: Change from the first in-person session to the second in person session of the intervention (2-weeks for Cohort 1 and 1-week for Cohort 2).
Population: Only those women who completed both of the in-person group sessions and provided complete data for the risk perception measure were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: number of key presses
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
Number analyzed (Participants) | 19 | 22
number of key presses | 6.58 (3.24) | 6.64 (8.98)
Statistical Analysis 1: Comparison: Revictimization Prevention for College Women (RPCW) vs Health Education Control (HEC); A one-way ANOVA was used to compare the mean difference in key presses from time 1 to time 2 between the intervention (RPCW) and Control conditions; Test type: Other; p < 0.99, ANOVA

4. Primary Outcome: Latency to Choose to Leave a Videotaped Scenario (Seconds)
Description: Time taken (Latency measured in seconds) to indicate a desire to leave a video depiction of a social interaction embedded with high-risk cues for sexual assault. Participants indicate when they are concerned about their sexual safety and would choose to exit the scenario if this were a live interaction by pressing a designated key on the computer keyboard (e.g., u). The measure is administered prior to and after the intervention and control condition, one week apart. A difference score (Time 2 - Time 1) is calculated. A reduced latency to choose to leave the scenario (i.e., choosing to leave more quickly) - indicates better recognition of risk.
Time Frame: as for outcome 3
Population: Individuals who had completed measure at both pre-intervention and post-intervention were included in analysis.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
Number analyzed (Participants) | 15 | 11
Seconds | -21.17 (23.36) | -6.34 (70.70)
Statistical Analysis 1: Comparison: Revictimization Prevention for College Women (RPCW) vs Health Education Control (HEC); Test type: Other; p < 0.45, ANOVA

5. Secondary Outcome: Difficulties in Emotion Regulation Scale
Description: Difficulties in Emotion Regulation Scale was used to assess emotion regulation; This scale consists of 36 items measured on a scale from 1 "almost never" to 5 "almost always." A higher score indicates greater ability to regulate emotions. Improvement would be an increase in score from time 1 to time 2.
  Minimum value is 36, Maximum value is 180. A higher score indicates a better outcome.
Time Frame: Assessed at baseline, 3-month follow up, and 6-month follow up (trait)
Population: Participants who completed the measure at all 3 time points were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
Number analyzed (Participants) | 27 | 18
score on a scale
  Baseline | 92.44 (28.59) | 87.39 (15.26)
  3-month Follow-up | 82.89 (26.95) | 83.61 (18.70)
  6-month Follow-up | 81.33 (24.97) | 82.72 (19.74)
Statistical Analysis 1: Comparison: Revictimization Prevention for College Women (RPCW) vs Health Education Control (HEC); Test type: Other; p < .10, ANOVA — Given the exploratory nature of the analysis we were looking for a trend in improvement in emotion regulation (i.e., p<.10) following the intervention condition compared to control

6. Secondary Outcome: State Difficulties in Emotion Regulation Scale
Description: Improvement in ability to regulate state emotion regulation as assessed by the State Difficulties in Emotion Regulation Scale; This scale consists of 21 items measured on a scale from 1 "not at all" to 5 "completely." A higher score is better, indicating greater ability to regulate emotions. Improvement in ability to regulate emotions is indicated by an increase in total score (summed score of all items, items on the awareness subscale are reverse coded before summing) from one time point to the next. Minimum score is 21, Maximum score is 105.
  A higher score means a better outcome.
Time Frame: as for outcome 3
Population: Participants who had complete data for both in-person group sessions. The state ders was administered prior to beginning the first in-person session (i.e., pre-intervention) and at the end of the second session (i.e, post-intervention).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
Number analyzed (Participants) | 28 | 28
score on a scale
  Pre-intervention | 38.57 (10.55) | 38.71 (11.04)
  Post-intervention | 35.79 (11.49) | 38.04 (10.6)
Statistical Analysis 1: Comparison: Revictimization Prevention for College Women (RPCW) vs Health Education Control (HEC); Repeated measure ANOVA was used to provide preliminary information for estimating sample sizes needed for a larger Stage II efficacy trial. The current pilot RCT was not powered to find significant effects; Test type: Other; p < .10, ANOVA

7. Secondary Outcome: The Protective Behavioral Strategies Scale
Description: The Protective Behavioral Strategies Scale (PBSS; 15-items; Martens et al., 2005; 2007) was used to assess use of drinking protective behavioral strategies. Each item is scored on frequency of use from 1 'never' to 6 'always' and summed for a total score, with higher scores indicating better use of drinking protective behavior strategies.
  Minimum value is 15, Maximum value is 90. Higher scores indicate a better outcome.
Time Frame: Assessed from baseline to the post-intervention survey; From post-intervention to the 3-month follow up; From 3- to 6-month follow up
Population: Participants who had data for all time points were included in the repeated measures ANOVA.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
Number analyzed (Participants) | 26 | 19
score on a scale
  Baseline | 58.23 (10.08) | 55.21 (10.91)
  Post-Intervention | 61.08 (10.21) | 60.00 (13.84)
  3-Month Follow-up | 61.92 (13.39) | 62.58 (12.83)
  6-Month Follow-up | 60.92 (11.73) | 61.53 (12.69)
Statistical Analysis 1: Comparison: Revictimization Prevention for College Women (RPCW) vs Health Education Control (HEC); An exploratory repeated measures ANOVA with time (4) as the within-subjects variable and condition (2) as the between-subjects variable was conducted to provide preliminary information for estimating sample sizes needed for a larger Stage II efficacy trial. The current pilot RCT was not powered to find significant effects; Test type: Other; p < .10, ANOVA — A priori threshold for a trend set at p<.10 for condition effect (intervention v control)

8. Secondary Outcome: The Dating Self-Protection Against Rape Scale
Description: The Dating Self-Protection against Rape Scale (DSPARS; Moore & Waterman, 1999; Scaglione et al., 2015) was used to assess 15 dating protective strategies. Each item is assessed using a 7-point scale from 1 "Never" to 7 "Always." A lower score is better, indicating less risky dating behavior. Minimum score is 15, maximum score is 105.
  Lower scores mean better outcome.
Time Frame: Assessed at baseline, post-intervention, 3-month follow up, and 6-month follow up
Population: Analysis included those participants who had complete data on the Dating Behavior Survey at all 4 time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
Number analyzed (Participants) | 26 | 18
score on a scale
  Baseline | 50.15 (8.15) | 55.61 (14.50)
  Post-intervention | 46.23 (8.20) | 52.67 (9.91)
  3-month follow-up | 49.65 (8.90) | 49.39 (8.77)
  6-month follow-up | 47.77 (7.08) | 51.50 (8.05)
Statistical Analysis 1: Comparison: Revictimization Prevention for College Women (RPCW) vs Health Education Control (HEC); An exploratory repeated measures ANOVA with time (4) as the within-subjects variable and condition (2) as the between-subjects variable was conducted to provide preliminary information for estimating sample sizes needed for a larger Stage II efficacy trial; Test type: Other; p < .098, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were assessed over the duration of the study from baseline through 6-month follow-up assessment (an average of 6 months) for each participant.
Description: clinicaltrials.gov definitions were used.
Arm/Group | Revictimization Prevention for College Women (RPCW) | Health Education Control (HEC)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 0/37 | 0/35

LIMITATIONS AND CAVEATS:
Although 90 women were eligible for the study, only 72 started the randomized control trial (RCT) and attrition after 6 months was higher than expected, reducing power for detecting significant differences in primary outcomes between the intervention and control groups. Given the pilot nature of the RCT and the good acceptability and feasibility of the intervention, slight modifications to the recruitment and retention procedures are likely to produce better efficacy in a larger RCT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT05257603/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05257603/SAP_001.pdf
  • Informed Consent Form (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT05257603/ICF_002.pdf